CLINICAL TRIAL: NCT01822379
Title: Comparative Study of the Use of Trypsin Versus Dispase in Melanocyte-Keratinocyte Transplantation for the Treatment of Vitiligo
Brief Title: Comparative Study of Techniques in Melanocyte-Keratinocyte Transplantation for the Treatment of Vitiligo
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This study was never initiated.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Senior Staff Physician, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB #6121
Record Dates: First submitted 2010-05-12; First posted 2013-04-02 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: diaspase versus trypsin for cell separation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Will perform cell separation using either diaspase or trypsin
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cell transplantation (Experimental): All patients will undergo transplantation of two distinct vitiligo lesions. One lesion will receive cells prepared with trypsin. The other lesion will receive cells prepared with dispase.
  Interventions: Procedure: Melanocyte Keratinocyte transplantation

INTERVENTIONS:
Procedure: Melanocyte Keratinocyte transplantation — Transplantation of cells prepared with dispase

SUMMARY:
Previous studies have evaluated the transplantation of pigment cells (melanocytes)and skin cells (keratinocytes) for the treatment of vitiligo. This procedure is known as MKTP (Melanocyte Keratinocyte Transplantation Procedure). Multiple studies have found this procedure to be both safe and effective for the treatment of vitiligo. The majority of these studies utilized trypsin to help isolate melanocytes and keratinocytes. Trypsin is enzyme that helps to separate the different layers of skin. However, some cell biologists believe that the enzyme dispase (which can be used to separate the epidermis from the dermis) is less toxic to cells of the epidermis and can result in a greater number of viable melanocytes and keratinocytes for transplantation.

This study will look at the repigmentation rates of MKTP using trypsin to isolate cells, versus MKTP using dispase to isolate cells.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old
2. Have a diagnosis of generalized vitiligo-vitiligo affecting both sides of the body on one or more areas of the body (extremities, trunk, etc.)
3. Have stable vitiligo, defined as no new lesion development (or expansion of existing lesions) in the 6 months prior to proposed procedure date
4. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form
5. Agree to follow and undergo all study-related procedures

Exclusion Criteria:

1. Female patients self-reported to be lactating, pregnant, or planning to become pregnant
2. Patients with a history of developing vitiligo or hypertrophic scars at sites of trauma
3. Patients self-reported as having HIV or Hepatitis C
4. Patients self-reported as having uncontrolled Diabetes Mellitus
5. The investigator feels the patient should not participate in the study for any reason
6. Patients with acral vitiligo, defined as significant involvement of the fingers and/or toes
7. Patients with focal or segmental vitiligo, defined as vitiligo affecting only one area of the body on only one side of the body
8. Patients with vitiligo affecting greater than 30% of their body surface area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pigmentation | 6 months
  Investigator will assess amount of pigmentation at site of procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H Hamzavi, MD, Principal Investigator — Henry Ford Dermatology
Locations (1):
- Henry Ford Hospital Department of Dermatology, Detroit, Michigan, United States